CLINICAL TRIAL: NCT00131105
Title: Combining Exercise and Diet in Older Adults
Brief Title: The TLC2 (Teaching Healthy Lifestyles to Caregivers 2)/CALM (Counseling Advice for Lifestyle Management) Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG0034; R01AG021010 (NIH)
Record Dates: First submitted 2005-08-15; First posted 2005-08-17 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Health Behavior; Psychological Stress; Healthy
Keywords: Healthy; Caregivers; Aging
MeSH Terms: conditions — Health Behavior; Stress, Psychological

INTERVENTIONS:
Behavioral: The Stanford Active Choices program

SUMMARY:
The purpose of this study is to evaluate the effects of a 12-month telephone-supervised, home-based physical activity and dietary intervention, conducted in either a sequential or simultaneous fashion, on improving physical activity and dietary patterns in a high-stress population.

DETAILED DESCRIPTION:
This study combines elements of two previous studies--Teaching Healthy Lifestyles for Caregivers (TLC2) and Counseling Advice for Lifestyle Management (CALM)--to compare exercise and diet interventions in caregivers and non-caregivers. Two hundred and forty healthy men and women ages 50 and older, half caregivers and half non-caregivers, will be randomly assigned to one of four conditions:

* a 12-month physical activity intervention and a 12-month dietary counseling intervention delivered simultaneously;
* a 12-month counseling intervention first focusing on physical activity followed by the addition of dietary counseling;
* a 12-month counseling intervention first focusing on dietary counseling followed by the addition of physical activity counseling; or
* a 12-month attention-control condition focusing on stress-management skills training.

Data on physical activity participation, saturated fat consumption, and related quality of life indicators (e.g., improved physical functioning, fitness, sleep, and psychological well-being) will be collected at baseline, 4 months, 8 months, and 12 months post-test. The primary hypotheses are:

* participants assigned to the physical activity and dietary counseling conditions will show greater improvements in physical activity participation and saturated fat consumption at 12 months compared to the attention-control condition; and
* participants in the sequentially-delivered counseling interventions will show greater improvements in physical activity and saturated fat consumption compared to participants in the simultaneously-delivered interventions.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 50 and older
* Current family caregiver
* Currently experiencing significant psychological stress
* Free of any medical condition that would limit participation in independent exercise
* Not currently engaged in a regular pattern of physical conditioning
* Current dietary pattern includes suboptimal total fat, saturated fat and vegetable and fruit consumption
* Free of chronic clinical psychopathology
* Stable on current medications
* Planning to remain in the geographic area throughout the duration of the trial
* Able to read and speak English sufficiently to understand protocol materials
* Able to use the telephone unaided
* Willing to accept random assignment to any study condition

Exclusion Criteria:

* Under the age of 50
* Currently under treatment for an acute, serious medical condition (e.g. cancer, heart disease, stroke)
* Physically active on a regular basis (i.e. performing more than 60 minutes per week of aerobic physical activity of at least a moderate intensity)
* Dietary patterns meet current recommendations for saturated fat and vegetable and fruit consumption
* Unstable and/or uncontrolled on medications for chronic medical conditions
* Unable or unwilling to use a telephone unaided
* Unwilling to accept random assignment to study condition

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2003-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Increase in aerobic physical activity measured by the Stanford 7-Day Physical Activity Recall | baseline, 4 months, 8 months, and 12 months
decrease in saturated fat measured by the Block food frequency questionnaire | baseline, 4 months, 8 months, and 12 months

SECONDARY OUTCOMES:
Physical performance on a symptom-limited, graded exercise treadmill test | baseline, 4 months, 8 months, and 12 months
quality of life and psychological questionnaires measuring physical functioning | baseline, 4 months, 8 months, and 12 months
sleep | baseline, 4 months, 8 months, and 12 months
perceived stress | baseline, 4 months, 8 months, and 12 months
depressive symptoms | baseline, 4 months, 8 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Abby C. King, PhD, Principal Investigator — Stanford Prevention Research Center
Locations (1):
- Stanford Prevention Research Center, Stanford, California, United States

REFERENCES:
- [Background] Wilcox S, King AC, Castro C, Bortz W. Do changes in physical activity lead to dietary changes in middle and old age? Am J Prev Med. 2000 May;18(4):276-83. doi: 10.1016/s0749-3797(00)00117-3. PMID 10788729
- [Background] King AC, Baumann K, O'Sullivan P, Wilcox S, Castro C. Effects of moderate-intensity exercise on physiological, behavioral, and emotional responses to family caregiving: a randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2002 Jan;57(1):M26-36. doi: 10.1093/gerona/57.1.m26. PMID 11773209
- [Background] Castro CM, Wilcox S, O'Sullivan P, Baumann K, King AC. An exercise program for women who are caring for relatives with dementia. Psychosom Med. 2002 May-Jun;64(3):458-68. doi: 10.1097/00006842-200205000-00010. PMID 12021419
- [Derived] Patel ML, Rodriguez Espinosa P, King AC. Moderators of a Diet and Physical Activity Intervention: who Responds Best to Sequential vs. Simultaneous Approaches. Int J Behav Med. 2025 Feb;32(1):80-91. doi: 10.1007/s12529-023-10223-9. Epub 2023 Oct 10. PMID 37816943
- [Derived] King AC, Castro CM, Buman MP, Hekler EB, Urizar GG Jr, Ahn DK. Behavioral impacts of sequentially versus simultaneously delivered dietary plus physical activity interventions: the CALM trial. Ann Behav Med. 2013 Oct;46(2):157-68. doi: 10.1007/s12160-013-9501-y. PMID 23609341